CLINICAL TRIAL: NCT06587620
Title: Tranexamic Acid Versus Dexmedetomidine for Improving Surgical Field Quality During Spine Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, manal mohamed rashad, Lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 11228-8/10-2023
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Surgical Field Quality Improvement in Spine Surgeries
MeSH Terms: interventions — Tranexamic Acid; Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (group c ) : saline (Placebo Comparator): IV infusion of 50 ml saline over 10 min before induction of anesthesia. IV saline infusion immediately after induction till 15 min before the end of surgery.
  Interventions: Other: Saline (NaCl 0,9 %) (placebo)
- Tranexamic acid group (group T) (Active Comparator): Start IV infusion of a loading dose of tranexamic acid 10 mg/kg completed to 50 ml saline over 10 min before induction of anesthesia. IV infusion of tranexamic acid at a dose of 1 mg/kg/h immediately after induction till 15 min before the end of surgery.
  Interventions: Drug: Tranexamic acid
- Dexmedetomidine group (group D). (Active Comparator): Start IV infusion of a loading dose of dexmedetomidine 1ug/kg completed to 50 ml saline over 10 min before induction of anesthesia. IV infusion of dexmedetomidine 0.3-0.7 µg/kg/h immediately after induction to maintain Mean Arterial Pressure (MAP) between 60-70 mmHg till 15 min before the end of surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Tranexamic acid — Start IV infusion of a loading dose of tranexamic acid 10 mg/kg completed to 50 ml saline over 10 min before induction of anesthesia. IV infusion of tranexamic acid at a dose of 1 mg/kg/h immediately after induction till 15 min before the end of surgery.
  Arms: Tranexamic acid group (group T)
Drug: Dexmedetomidine — Start IV infusion of a loading dose of dexmedetomidine 1ug/kg completed to 50 ml saline over 10 min before induction of anesthesia. IV infusion of dexmedetomidine 0.3-0.7 µg/kg/h immediately after induction to maintain Mean Arterial Pressure (MAP) between 60-70 mmHg till 15 min before the end of surgery.
  Arms: Dexmedetomidine group (group D).
Other: Saline (NaCl 0,9 %) (placebo) — IV infusion of 50 ml saline over 10 min before induction of anesthesia. IV saline infusion immediately after induction till 15 min before the end of surgery.
  Arms: control group (group c ) : saline

SUMMARY:
The most common procedure said to involve substantial bleeding is spine surgery. There is always a significant danger of bleeding and blood transfusion associated with these procedures, particularly complex and multilevel spine surgeries. Care of bleeding should be taken, as excessive blood loss can lead to impaired vision of surgical field, anemia, postoperative epidural hematoma and transfusion-related complications as transfusion reactions and transmission of infections.

For these reasons, improving surgical field is a must. Hemostasis procedures, including good positioning, controlled hypotension, local vasoconstrictors, epidural block, biological and chemical medications including desmopressin, aprotinin, tranexamic acid, epsilon, aminocaproic acid, dexmedetomidine, can all be used to decrease bleeding.

and In this study we compared the effect of tranexamic acid and dexmedetomidine on hemodynamics, blood loss, transfusion and the quality of the surgical field.

Sample size was 78 cases who underwent lumbar decompression and fixation surgery at 2 levels. They were divided into 3 equal groups (26 patients in each one) :

1. Control grup (group C): received loading IV infusion of 50 ml saline over 10 min before induction of anesthesia, then maintenance IV infusion of saline.
2. Tranexamic acid group (group T): received loading dose of tranexamic acid 10 mg/kg over 10 min before induction of

   anesthesia, then maintenance IV infusion of tranexamic acid 1mg/kg/h.
3. Dexmedetomidine group (group D): received loading dose of dexmedetomidine 1 μg/kg over 10 min before induction of anesthesia, then maintenance IV infusion of dexmedetomidine 0.3-0.7 μg/kg/h.

We compared the 3 groups regarding these characteristics : - Age, sex, body mass index and ASA classification

* Hemodynamics (mean arterial pressure & heart rate) and oxygen saturation.
* Amount of blood loss, blood transfusion, pre and post operative hemoglobin and hematocrit levels.
* Side effects, duration of surgery, emergence and discharge times.
* Score of intraoperative surgical field. The results revealed that dexmedetomidine achieved more hypotensive and bradycardiac effects than other study drugs, but tranexamic acid had the upper hand in decreasing the amount of blood loss and blood transfusion. Side effects were more in dexmedetomidine group than other groups, represented mainly as hypotension and bradycardia. Duration of surgery was shorter in tranexamic acid group than other groups. Emergence and discharge times were longer in dexmedetomidine group than other groups. There was no statistical significant difference between the 3 groups in surgical field score.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent. 2. Age: 21-60 years old. 3. Physical status: ASA І & II. 4. BMI: 18.5-30 kg/m2. 5. Type of operations : elective lumbar decompression and fixation surgeries at 2 levels. 6. Time of operation : less than 4 hours. 7. Type of anesthesia : general anesthesia.

Exclusion Criteria:

* 1. known history of allergy to study drugs. 2. Central nervous system disorder and metabolic diseases. 3. History or risk of thrombosis or active thromboembolic disease as deep vein thrombosis and pulmonary embolism. 4. Coagulopathies or taking drugs affecting coagulation ( INR>1.5 , PLatelets count less than 100.000 per microliter of blood ). 5. Patients on B- blockers.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The effect of tranexamic acid and dexmedetomidine on improving surgical field quality | 240 minuets
  The visibility of the surgical field was assessed by surgeon using Boezaart scoring system throughout the operation

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of medicine, zagazig university, Zagazig, Elsharqya
  - Zagazig University, Zagazig

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoo JS, Ahn J, Karmarkar SS, Lamoutte EH, Singh K. The use of tranexamic acid in spine surgery. Ann Transl Med. 2019 Sep;7(Suppl 5):S172. doi: 10.21037/atm.2019.05.36. PMID 31624738
- [Background] Tasbihgou SR, Barends CRM, Absalom AR. The role of dexmedetomidine in neurosurgery. Best Pract Res Clin Anaesthesiol. 2021 Jul;35(2):221-229. doi: 10.1016/j.bpa.2020.10.002. Epub 2020 Oct 14. PMID 34030806
- [Background] Ruku R, Jamwal A, Bhadrala N, Gulati S. Randomized Open-Labelled Comparative Evaluation of the Efficacy of Nitroglycerine, Esmolol and Dexmedetomidine in Producing Controlled Hypotension in Spine Surgeries. Anesth Essays Res. 2019 Jul-Sep;13(3):486-491. doi: 10.4103/aer.AER_78_19. PMID 31602066
- [Background] Kundra S, Taneja S, Choudhary AK, Katyal S, Garg I, Roy R. Effect of a low-dose dexmedetomidine infusion on intraoperative hemodynamics, anesthetic requirements and recovery profile in patients undergoing lumbar spine surgery. J Anaesthesiol Clin Pharmacol. 2019 Apr-Jun;35(2):248-253. doi: 10.4103/joacp.JOACP_338_18. PMID 31303717
- [Background] Ahmadi MS, Jahanshahi J, Hashemian F, Salimbahrani AR, Haghi N, Khanlarzadeh E. Comparison of Tranexamic Acid and Dexmedetomidine on Bleeding in Endoscopic Sinus Surgery. Iran J Otorhinolaryngol. 2023 Jan;35(126):49-56. doi: 10.22038/IJORL.2022.64361.3203. PMID 36721414
- [Background] Modir H, Moshiri E, Naseri N, Faraji F, Almasi-Hashiani A. A randomized parallel design trial of the efficacy and safety of tranexamic acid, dexmedetomidine and nitroglycerin in controlling intraoperative bleeding and improving surgical field quality during septorhinoplasty under general anesthesia. Med Gas Res. 2021 Oct-Dec;11(4):131-137. doi: 10.4103/2045-9912.318857. PMID 34213494